CLINICAL TRIAL: NCT04853953
Title: Incidence of Bleeding Complications in Critically Ill COVID-19 Patients With Acute Respiratory Distress Syndrome on Veno-venous ECMO
Brief Title: Cerebral Bleeding in COVID-19 ARDS Patients on Veno-venous ECMO
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Zurich (Other)
Collaborators: Hannover Medical School (Other); University Hospital, Bonn (Other)
Responsible Party: Sponsor
Other Study IDs: SD03
Record Dates: First submitted 2021-04-16; First posted 2021-04-22 (Actual); Last update posted 2021-04-22 (Actual); Status verified 2021-04

CONDITIONS: Acute Respiratory Distress Syndrome; Extracorporeal Membrane Oxygenation Complication; Corona Virus Infection
MeSH Terms: conditions — Respiratory Distress Syndrome; Coronavirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COVID-19 ARDS patients requiring veno-venous ECMO support: Critically ill COVID-19 patients with ARDS requiring ECMO support will be analyzed in this group. Patients from all three study sites will be assessed for participation.
  Interventions: Other: Incidence of bleeding complications in ARDS patients on veno-venous ECMO
- Non-COVID-19 ARDS patients requiring veno-venous ECMO support: Critically ill Non-COVID-19 patients with ARDS requiring ECMO support will be analyzed in this group. Patients from all three study sites will be assessed for participation.
  Interventions: Other: Incidence of bleeding complications in ARDS patients on veno-venous ECMO

INTERVENTIONS:
Other: Incidence of bleeding complications in ARDS patients on veno-venous ECMO — All bleeding complications (especially cerebral bleedings) will be analyzed in the study groups. At the bleeding event, laboratory parameters of coagulation will be collected and the intensity of the ECMO treatment

SUMMARY:
Critically ill patients with severe acute respiratory distress syndrome (ARDS) sometimes require treatment with veno-venous extracorporeal membrane oxygenation (ECMO) to support gas exchange. To prevent clotting of the ECMO circuit, these patients need to be anticoagulated. This protective anticoagulation also leeds to an increased bleeding risk.

Most critically ill COVID-19 patients suffer from an ARDS and some require ECMO support. However, the optimal strategy and targets for the anticoagulation of these patients remain uncertain. Studies have shown that COVID-19 is associated with endotheliopathy probably leading to procoagulatory effects. On the other hand, the incidence of bleeding complications associated with this endotheliopathy is not clear and remains to be elucidated.

Anticoagulation of COVID-19 patients on ECMO thus poses a challenge for clinicians.

The hypothesis of the current project is that COVID-19 patients with ARDS on ECMO exhibit a higher number of bleeding complications compared to historical control patients with non-COVID-19 ARDS requiring ECMO support.

DETAILED DESCRIPTION:
The primary aim of the project is to retrospectively analyze the incidence of bleeding complications (especially cerebral bleedings) in critically ill COVID-19 patients with ARDS requiring ECMO support. The incidences of bleeding will be compared with a historical control cohort of non-COVID-19 patients on ECMO support.

The data analysis will be set up within a multicentric, retrospective study involving the University Hospital Zurich (Switzerland), the Medical School Hannover (Germany) and the University Hospital Bonn (Germany). The aim of the multicentric approach is to increase the case load and to improve the validity of the data, which could possibly have therapeutic implications in the future.

Aside from demographic and baseline date, mortality and causes of death, comorbidities, the anticoagulation strategy (substance, targets of anticoagulation) and laboratory parameters of the anticoagulation during the bleeding events will be collected.

Furthermore, the intensity of the ECMO treatment (blood flow, sweep gas flow, oxygen requirement) during the bleeding events and the catecholamine use during ECMO implantation will be analyzed.

To enhance comparability, intensive care specific treatments (proning, sedation and analgesia, COVID-19 targeted therapy) will be collected and analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Critically ill patients with ARDS requiring ECMO support from all three study sites
* age > 18 years

Exclusion Criteria:

- Presence of an objective, declared denial to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of critically ill COVID-19 and Non-COVID-19 ARDS patients requiring veno-venous ECMO support.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2021-04-30 (Estimated); Primary Completion 2021-07 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Cerebral bleedings in critically ill ARDS patients requiring ECMO support | From date of inclusion of patients into the study, all outcome measures will be analyzed in a time-to-event analysis ranging from ICU admission up to the bleeding event, assessed up to six months
  Cerebral bleedings will be analyzed and classified according to cerebral imaging (computed tomography, magnetic resonance tomography)

SECONDARY OUTCOMES:
Non-cerebral bleedings in critically ill ARDS patients requiring ECMO support | From date of inclusion of patients into the study, all outcome measures will be analyzed in a time-to-event analysis ranging from ICU admission up to the bleeding event, assessed up to six months
  Bleedings will be classified according to the documentation in the electronic medical reports

CONTACTS AND LOCATIONS:
Overall Officials: Sascha David, Prof, Principal Investigator — University Hospital Zurich, Institute of Intensive Care

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Makdisi G, Wang IW. Extra Corporeal Membrane Oxygenation (ECMO) review of a lifesaving technology. J Thorac Dis. 2015 Jul;7(7):E166-76. doi: 10.3978/j.issn.2072-1439.2015.07.17. PMID 26380745
- [Result] Rawal G, Yadav S, Kumar R. Acute Respiratory Distress Syndrome: An Update and Review. J Transl Int Med. 2018 Jun 26;6(2):74-77. doi: 10.1515/jtim-2016-0012. eCollection 2018 Jun. PMID 29984201
- [Result] Varga Z, Flammer AJ, Steiger P, Haberecker M, Andermatt R, Zinkernagel AS, Mehra MR, Schuepbach RA, Ruschitzka F, Moch H. Endothelial cell infection and endotheliitis in COVID-19. Lancet. 2020 May 2;395(10234):1417-1418. doi: 10.1016/S0140-6736(20)30937-5. Epub 2020 Apr 21. No abstract available. PMID 32325026
- [Derived] Seeliger B, Doebler M, Hofmaenner DA, Wendel-Garcia PD, Schuepbach RA, Schmidt JJ, Welte T, Hoeper MM, Gillmann HJ, Kuehn C, Ehrentraut SF, Schewe JC, Putensen C, Stahl K, Bode C, David S. Intracranial Hemorrhages on Extracorporeal Membrane Oxygenation: Differences Between COVID-19 and Other Viral Acute Respiratory Distress Syndrome. Crit Care Med. 2022 Jun 1;50(6):e526-e538. doi: 10.1097/CCM.0000000000005441. Epub 2022 Jan 12. PMID 35020672